CLINICAL TRIAL: NCT02631512
Title: Evaluation of Woulgan in Diabetic Foot Ulcer Compared With a Commercial Hydrogel
Brief Title: Evaluation of Woulgan in Diabetic Foot Ulcer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotec Pharmacon ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WBG-03
Record Dates: First submitted 2015-11-09; First posted 2015-12-16 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Woulgan Gel (Other): Primary dressing with Woulgan Gel with Soluble Beta-Glucan (SBG)
  Interventions: Device: Woulgan Gel
- Intrasite Hydrogel (Other): Primary dressing with Intrasite Hydrogel
  Interventions: Device: Intrasite Hydrogel

INTERVENTIONS:
Device: Woulgan Gel — Primary dressing gel to be applied to the wound bed, and to be covered with a secondary bandage.
  Arms: Woulgan Gel
Device: Intrasite Hydrogel — Primary dressing hydrogel to be applied to the wound bed, and to be covered with a secondary bandage
  Arms: Intrasite Hydrogel

SUMMARY:
The aim of the current study is to support the performance and safety of Woulgan® in the treatment of diabetic foot ulcer in comparison with the commercially available hydrogel Intrasite. Healing and untoward medical events to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type I or II diabetes mellitus.
* Target ulcer area between 0.5 and 5 sqcm, and more than 4 weeks old.
* Ankle-brachial pressure index above 0.7.

Exclusion Criteria:

* Ulcers due to non-diabetic etiology.
* Uncontrolled diabetes defined as HbA1c above 70 mmol/mol and insufficient nutritional status.
* Ulcers older than 1 year.
* Any of gangrene, osteomyelitis, cellulitis, or Charcot osteoarthropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Performance of Woulgan Gel as primary dressing in diabetic foot ulcer in terms of reduced wound size in sqcm. | Until 8 weeks from start of treatment

SECONDARY OUTCOMES:
Safety of Woulgan Gel as primary dressing in diabetic foot ulcer measured in terms of untoward medical events | Until 8 weeks from start of treatment
Useability of Woulgan as primary dressing in diabetic foot ulcer measured as degree of pain (100 mm VAS). | Until 8 weeks from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Londahl, MD, PhD, Principal Investigator — Skane University Hospital
Locations (3):
- Skaane University Hospital, Lund, Sweden
- United Kingdom (2):
  - North Middlesex University Hospital, London
  - Nottingham University Hospital, Nottingham